CLINICAL TRIAL: NCT00092105
Title: A Multicenter, Double-Blind, Randomized, Crossover Study Investigating the Clinical Effect of Montelukast in Patients With Concomitant Asthma and Allergic Rhinitis Upon Controlled Exposure to Cat Allergen
Brief Title: Study of MK0476 (Montelukast Sodium) and Effects on Asthma and Nasal Symptoms Upon Exposure to Cats (0476-256)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 0476-256; 2004_024
Record Dates: First submitted 2004-09-21; First posted 2004-09-24 (Estimated); Last update posted 2024-08-14 (Actual); Status verified 2022-02

CONDITIONS: Asthma, Bronchial; Rhinitis, Allergic, Perennial
Keywords: Rhinitis, Allergic
MeSH Terms: conditions — Asthma; Rhinitis, Allergic, Perennial; Rhinitis, Allergic | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0476, montelukast sodium
Drug: Comparator: placebo

SUMMARY:
The purpose of this study is to determine the protective effect of an approved medication on asthma and allergic rhinitis (inflammation of the mucous membrane of the nose) upon exposure to cats.

DETAILED DESCRIPTION:
The duration of treatment is 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Increased sensitivity to cat allergen proven by positive allergy testing, and by decreased lung function and increased symptoms of allergic rhinitis (runny nose) upon exposure to cats.

Exclusion Criteria:

* Medical history of a lung disorder (other than asthma) or a recent upper respiratory tract infection.

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2002-04-01 (Actual); Primary Completion 2003-01-01 (Actual); Study Completion 2003-01-28 (Actual)

PRIMARY OUTCOMES:
Co-Primary endpoints: (1) Area Under the Curve (AUC) for the percent fall from prechallenge FEV1 during allergen challenge; (2) Area Under the Curve for the increase from prechallenge Nasal Symptoms score during allergen challenge

SECONDARY OUTCOMES:
(1) Maximum percent fall from prechallenge FEV1; (2) AUC for the increase from prechallenge Chest Symptoms score (3) AUC for the increase from prechallenge Nasal Symptoms score collected over 60 minutes after terminating the challenge.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Perry TT, Corren J, Philip G, Kim EH, Conover-Walker MK, Malice MP, Massaad R, Dass SB, Reiss TF, Wood RA. Protective effect of montelukast on lower and upper respiratory tract responses to short-term cat allergen exposure. Ann Allergy Asthma Immunol. 2004 Nov;93(5):431-8. doi: 10.1016/S1081-1206(10)61409-3. PMID 15562881